CLINICAL TRIAL: NCT05412940
Title: Accelerometry and Rehabilitation After Knee Replacement Study (ARK): A Prospective, Randomised Controlled Trial.
Brief Title: Accelerometry and Rehabilitation After Knee Replacement Study (ARK)
Acronym: ARK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OR21/144310
Record Dates: First submitted 2022-01-21; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary total knee replacement patients

SUMMARY:
Total knee replacement (TKR) is a successful and cost-effective treatment for end-stage arthritis. Its usage is increasing due to changing population demographics and quality of life (QoL) expectations. There were almost 100,000 total knee replacements (TKR) performed in England between 2018/19. After TKR, patient engagement in their rehabilitation exercises is very important but physiotherapy services are very stretched at present especially in the covid-19 era. Patient compliance with their exercises is poor at about 25%.

The use of wearable sensors (WS) following TKR is gaining lots of interest especially in the post covid-era. A recent review found five small studies which supported the feasibility of their use. WS may help with patients to engage better with their rehabilitation exercises after surgery, delivering remote physiotherapy and potentially help identify patients who may be struggling more and therefore need further targeted help with physiotherapy.

Sensors have the potential to be a cost-saving intervention for the NHS by improving efficiencies in monitoring patients by reducing number of outpatient appointments, reducing rehabilitation time, improving patient's adherence to rehabilitation schedules and increasing confidence in exercise regimes leading to improved health-related quality of life. We will conduct the first large scale study where 250 patients having TKR will be randomly chosen to either receive a WS (125 patients) against 125 patients who will have standard care (SC). Patient reported outcomes (PROMs), pain scores, objective measures of knee function and data from the sensors on how well patients engaged with their exercises will be collected. The study will also assess if WS is cost effective, at 6 months after surgery.

This study has the potential to revolutionise how pre- and post-knee replacement rehabilitation is delivered, providing an individualised, cost effective and successful solution to the current status.

ELIGIBILITY:
Inclusion Criteria:

* • Primary total knee replacement patients

  * Participant is aged 18 years of age or over
  * Participant is able and willing to provide written informed consent
  * Participant with ability to work with smart devices
  * Participant having own device (Apple iPhone or iPad or Android tablet or smartphone - minimum requirement: IOS - 12.4 or later/Android - 6.5 or later)
  * Internet connection at patient's home - either Wifi or mobile internet (min. 3G)

Exclusion Criteria:

* • Participants who are unwilling or mentally and/or physically unable to adhere to study procedures

  * Participants with dementia or other cognitive impairment which would prevent them from using the sensor/app
  * Presence of a previous joint replacement in the same knee
  * Surgical treatment of involved knee within the past 6 months (excluding arthroscopy)
  * Previous orthopaedic surgery for trauma or arthritis of the knee joint (such as a previous fracture fixation or osteotomy)
  * Active cancer (currently diagnosed and under treatment)
  * Unable to complete all trial procedures (e.g. attend follow up visits, complete questionnaires)
  * Unable to provide informed consent (cognitive disorder such as dementia, psychiatric illness)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Operating lists will be screened by the clinical trials team to identify eligible patients and patient information sheets will be sent out with invitation to meet surgeon and confirm eligibility.
  2. Potentially eligible patients will be provided with a patient information sheet at their routine pre-operative outpatient clinic and their eligibility confirmed by their operating surgeon
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of Oxford Knee Score (OKS) at 6 months from surgery | 6 months
  Completion of Patient satisfaction at 6 months after surgery using a survey questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom